CLINICAL TRIAL: NCT05683574
Title: Parallel-Group,Double-Blind,Double-Dummy,Superiority Study of Etoricoxib90mg/ Cyclobenzaprine15mg From Eurofarma Versus Etoricoxib90mg (Arcoxia®) and Cyclobenzaprine15mg (XL - Mitrul®) for Muscle Spasm After Third Molar Extraction in Brazil
Brief Title: Fixed-dose Combination of Etoricoxib + Cyclobenzaprine for Pain Relief After Third Molar Extraction in Brazil
Acronym: BENCOX
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Change in study strategy.
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EF 181
Record Dates: First submitted 2022-12-01; First posted 2023-01-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Third Molar Extraction
MeSH Terms: interventions — cyclobenzaprine; Etoricoxib

STUDY DESIGN:
Intervention Model Description: Participants who meet all eligibility criteria will be randomized to one of the following treatment groups:
  Investigational group: FDC of etoricoxib 90 mg + cyclobenzaprine 15 mg from Eurofarma Laboratórios SA (investigational drug). Participants randomized to this group will receive one (01) capsule of the investigational drug when postoperative pain intensity reaches moderate to serious intensity (≥ 40 mm at VAS 0-100 mm) and one (01) etoricoxib placebo tablet. The participants will be instructed, from then on, to use this same treatment, respecting a minimum interval of twenty-four (24) hours between doses for 3 days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Comparator Group: etoricoxib 90 mg (Arcoxia®). Participants randomized to this group will receive one (01) etoricoxib 90 mg tablet (Arcoxia®) when postoperative pain intensity reaches moderate to serious intensity (≥ 40 mm at VAS 0-100 mm) and one (01) FDC placebo capsule. The participants will be instructed, from then on, to use this same treatment, respecting a minimum interval of twenty-four (24) hours between doses for 3 days.
  Comparator Group: cyclobenzaprine hydrochloride 15 mg (XL - Mitrul®). Participants randomized to this group will receive one (01) cyclobenzaprine hydrochloride 15 mg capsule (XL - Mitrul®) (which will be masked inside a capsule like the FDC) when postoperative pain intensity reaches moderate to serious intensity (≥ 40 mm at VAS 0-100 mm) and one (01) etoricoxib placebo tablet. The participants will be instructed, from then on, to use this same treatment, respecting a minimum interval of twenty-four (24) hours between doses for 3 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- etoricoxib 90 mg + cyclobenzaprine 15 mg (Experimental): Investigational group: FDC of etoricoxib 90 mg + cyclobenzaprine 15 mg from Eurofarma Laboratórios SA
  Interventions: Drug: FDC of etoricoxib + cyclobenzaprine + etoricoxib placebo
- etoricoxib 90 mg (Active Comparator): Comparator group: etoricoxib 90 mg (Arcoxia®)
  Interventions: Drug: etoricoxib 90 mg (Arcoxia®) +FDC placebo
- cyclobenzaprine hydrochloride 15 mg (Active Comparator): Comparator group: cyclobenzaprine hydrochloride 15 mg (XL - Mitrul®)
  Interventions: Drug: cyclobenzaprine hydrochloride + etoricoxib placebo

INTERVENTIONS:
Drug: FDC of etoricoxib + cyclobenzaprine + etoricoxib placebo — Participants randomized to this group will receive one (01) capsule of the investigational drug and one (01) etoricoxib placebo tablet, respecting a minimum interval of twenty-four (24) hours between doses for 3 days.
  Other Names: Investigation drug 1
  Arms: etoricoxib 90 mg + cyclobenzaprine 15 mg
Drug: etoricoxib 90 mg (Arcoxia®) +FDC placebo — Participants randomized to this group will receive one (01) etoricoxib 90 mg tablet (Arcoxia®) and one (01) FDC placebo capsule, respecting a minimum interval of twenty-four (24) hours between doses for 3 days.
  Other Names: Comparator drug 2
  Arms: etoricoxib 90 mg
Drug: cyclobenzaprine hydrochloride + etoricoxib placebo — Participants randomized to this group will receive one (01) cyclobenzaprine hydrochloride 15 mg capsule (XL - Mitrul®) and one (01) etoricoxib placebo tablet, respecting a minimum interval of twenty-four (24) hours between doses for 3 days.
  Other Names: Comparator drug 3
  Arms: cyclobenzaprine hydrochloride 15 mg

SUMMARY:
Etoricoxib and cyclobenzaprine hydrochloride are active pharmaceutical ingredients (APIs) already registered in the country as mono-drugs. These products are widely used for the proposed indications, and their safety and efficacy profiles are known in daily clinical practice. Once the absence of a pharmacokinetic interaction between etoricoxib and cyclobenzaprine hydrochloride has been confirmed in relative bioavailability studies, this phase 3 study will be conducted for demonstrating the superiority of the new FDC over etoricoxib 90 mg (Arcoxia®) and cyclobenzaprine hydrochloride 15 mg (XL - Mitrul®) in the treatment of moderate to serious pain associated with muscle spasm. The purpose is to provide a new, effective, and safe therapeutic option to address these cases. Etoricoxib and cyclobenzaprine hydrochloride are active pharmaceutical ingredients (APIs) already registered in the country as mono-drugs. These products are widely used for the proposed indications, and their safety and efficacy profiles are known in daily clinical practice. Once the absence of a pharmacokinetic interaction between etoricoxib and cyclobenzaprine hydrochloride has been confirmed in relative bioavailability studies, this phase 3 study will be conducted for demonstrating the superiority of the new FDC over etoricoxib 90 mg (Arcoxia®) and cyclobenzaprine hydrochloride 15 mg (XL - Mitrul®) in the treatment of moderate to serious pain associated with muscle spasm. The purpose is to provide a new, effective, and safe therapeutic option to address these cases.

DETAILED DESCRIPTION:
The investigational drug consists of a fixed-dose combination (FDC) that contains etoricoxib, a non-steroidal anti-inflammatory drug (NSAID) with analgesic action, and cyclobenzaprine hydrochloride, a myorelaxant, in doses of 90 mg and 15 mg, respectively, in the dosage form of a prolonged-release hard capsule. This product is an unprecedented FDC in the country, and is indicated for the short-term treatment of moderate to serious acute pain associated with muscle spasm. Pain management with analgesic drugs, such as NSAIDs and other adjuvant drugs, is common in daily clinical practice. In parallel with its additive effect on pain relief, the FDC of an anti-inflammatory and myorelaxant agent seeks to assist in greater control of associated musculoskeletal symptoms, such as inflammatory processes, limited range of motion, and muscle spasms.

Multicenter, Randomized, Parallel-Group, Double-Blind, Double-Dummy, Comparative Superiority clinical trial. Patients aged between 18 and 35 years with indication for surgical removal of an impacted lower third molar and an antagonistic upper third molar will be randomized in a 1:1:1 ratio to receive the FDC of etoricoxib 90 mg + cyclobenzaprine hydrochloride 15 mg from Eurofarma Laboratórios SA (investigational drug), in capsules, or the mono-drugs etoricoxib 90 mg (Arcoxia®), in tablets, or cyclobenzaprine hydrochloride 15 mg (XL - Mitrul®), in capsules, for up to three (03) days. Participants whose surgery lasts a maximum of 80 minutes (counted from the initial incision to the extraction of the third molars) and who present moderate to serious postoperative pain up to a maximum of four (04) hours will be randomized. The first administration of study treatment will be made at the study center when post-surgical pain reaches moderate/serious intensity (≥ 40 mm on visual analogue scale [VAS] 0-100 mm). The participants will be instructed, from then on, to use the study treatment, respecting a minimum interval of twenty-four (24) hours between doses taken for three (03) days.

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes who meet all of the following criteria will be included in the study:

* Age between 18 and 35 years (inclusive).
* Presence of at least one lower third molar with partial or total bone inclusion (occlusal surface partially or completely covered by bone tissue) with indication for surgical removal (diagnosis made by panoramic radiograph taken within the six [06] months prior to study enrollment), in a vertical, mesioangular or horizontal position according to the Winter classification1,provided they belong to the following Pell & Gregory classes2:

  * Impacted lower third molar in vertical or mesioangular position: may be included, as long as it belongs to Pell & Gregory classes Ia, Ib, IIa or IIb;
  * Lower third molar impacted in a horizontal position: may be included, as long as it belongs to Pell & Gregory classes Ia, Ib or IIa.

Exclusion Criteria:

Patients who meet at least one of the following criteria will be excluded from the study:

* Presence of previous inflammatory and/or infectious oral lesion with indication for the use of anti-inflammatory agent and/or antibiotic therapy.
* Presence of any oral lesion in the region of the third molar to be extracted that may contraindicate extraction, at the discretion of the dental team (for example, pericoronitis, periodontitis, cysts, among others).
* Smoking* *Any use of tobacco, including e-cigarettes, is prohibited during the study. In the case of the participant who occasionally smokes, he/she must be willing not to use tobacco throughout his/her participation in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2026-05-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy variable is composed of the sum of the scores for pain relief within 6 h | The primary efficacy variable is an endpoint composed of the sum of pain relief scores within 6 hours and the percentage of postoperative mouth opening.
  The primary efficacy variable is composed of the sum of the scores for pain relief within 6 hours and the percentage of postoperative mouth opening. After administration of the first dose, participants will rate pain relief on a 5-point categorical scale at hourly intervals (1 hour, 2 hours, 3 hours, 4 hours, 5 hours and 6 hours). Clinical success is defined as very relief (scale 3) or complete relief (scale 4) within 6 hours after treatment administration.
Primary Efficacy Endpoint - Mouth opening will be calculated from the average of three measurements | Clinical success in this variable is defined as a mouth opening ≥ 80% in relation to the preoperative period.
  Mouth opening will be calculated from the average of three measurements that will be taken twice at the randomization visit and at visit 1, the evaluation visit, after three days. The measurement will be made using a calibrated digital caliper, considering the distance between upper and lower central incisors. The percentage of mouth opening at the evaluation visit will be calculated in reference to the baseline opening observed at the randomization visit. Clinical success in this variable is defined as a mouth opening ≥ 80% compared to the preoperative period.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints - Proportion of patients reporting much relief or complete relief in TOTPAR question items within 6 hours | Proportion of patients reporting much relief or complete relief in TOTPAR question items within 6 hours.
  The two clinical success criteria, defined as components of the primary endpoint, will be described as secondary endpoints:
  Proportion of patients reporting much relief or complete relief in TOTPAR question items within 6 hours.
Secondary Efficacy Endpoints - Proportion of patients who maintained at least 80% of full mouth opening three days after the procedure | Proportion of patients who maintained at least 80% of full mouth opening three days after the procedure.
  Proportion of patients who maintained at least 80% of full mouth opening three days after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, São Paulo, Brazil